CLINICAL TRIAL: NCT02582827
Title: A Phase I Trial of ABI-011 Administered Weekly in Patients With Advanced Solid Tumors or Lymphomas
Brief Title: QUILT-3.014: A Trial of ABI-011 Administered Weekly in Patients With Advanced Solid Tumors or Lymphomas
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Enrollment not initiated
Sponsor: NantBioScience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-3.014
Record Dates: First submitted 2015-10-14; First posted 2015-10-21 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2018-09

CONDITIONS: Neoplastic Disease
Keywords: Advanced Solid Tumors; solid tumor; lymphoma
MeSH Terms: conditions — Neoplasms; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ABI-011 (Experimental): IDN 5404 protein-bound particles for injectable suspension
  Interventions: Drug: ABI-011

INTERVENTIONS:
Drug: ABI-011 — ABI-011 is a novel, albumin-bound formulation of a potent thiocolchicine analog, IDN 5404, with a mean particle size of approximately 100 nm.
  Other Names: IDN 5404 protein-bound particles for injectable suspension

SUMMARY:
The primary objective of study CA601.2 is to determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of ABI-011 when administered by intravenous (IV) infusion on Days 1, 8, and 15, followed by a week of rest, in patients with advanced solid tumor malignancies or lymphomas. The MTD will be determined using a standard 3+3 design. The secondary objectives are to evaluate the safety and toxicity profile, to evaluate the plasma pharmacokinetics (PK), to assess the biological activity and pharmacodynamics, and to make a preliminary assessment of tumor response in patients with advanced solid tumors or lymphomas. The exploratory objectives are to determine the genomic and proteomic profile of patients' tumors to identify gene mutations, gene amplifications, levels of protein expression, and pinpoint oncoproteins. Correlations between genomic/proteomic profiles and efficacy outcomes will be assessed and principal metabolites of ABI-011 will be determined, if possible.

Approximately 45-60 patients will be treated to determine dose limiting toxicities (DLTs), the MTD, and/or RP2D of ABI-011. Once the RP2D is identified, expansion of this cohort (up to 10 patients) will occur.

DETAILED DESCRIPTION:
ABI-011 is a novel, albumin-bound formulation of a potent thiocolchicine analog, IDN 5404, with a mean particle size of approximately 100 nanometers (nm). The active drug, IDN 5404, is related to the colchicine family of tubulin-binding compounds that have been found to have vascular-disrupting activity in vivo. Studies are ongoing to determine whether IDN 5404 has vascular-disrupting activity. As a dimer, IDN 5404 has an additional activity as an inhibitor of topoisomerase I, a critical enzyme in deoxyribonucleic acid (DNA) repair mechanisms. Although the active compound has limited solubility, IDN 5404 formulated as ABI-011 is soluble in saline, facilitating IV dosing and delivery of the active agent to tumors and the tumor vasculature.

The primary objective of study CA601.2 is to determine the MTD or RP2D of ABI-011 when administered by IV infusion on Days 1, 8, and 15, followed by a week of rest, in patients with advanced solid tumor malignancies or lymphomas. The MTD will be determined using a standard 3+3 design. The secondary objectives are to evaluate the safety and toxicity profile, to evaluate the plasma PK (elimination rate constant, elimination half-life, volume of distribution, maximum serum concentration (Cmax), time to maximum concentration (tmax), and area under the time-concentration curve to time infinity (AUCinf), to assess the biological activity and pharmacodynamics, and to make a preliminary assessment of tumor response in patients with advanced solid tumors or lymphomas. The exploratory objectives are to determine the genomic and proteomic profile of patients' tumors to identify gene mutations, gene amplifications, levels of protein expression, and pinpoint oncoproteins. Correlations between genomic/proteomic profiles and efficacy outcomes will be assessed and principal metabolites of ABI-011 will be determined, if possible.

Approximately 45-60 patients will be treated to determine DLTs, the MTD, and/or RP2D of ABI-011. Once the RP2D is identified, expansion of this cohort (up to 10 patients) will occur.

Patients with cytologically or histologically confirmed solid tumor malignancies or lymphoma for which no curative standard approved therapy is available with an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 will be included. In the dose-escalation phase of the study, patients can have measurable or non-measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1, criteria. In the dose-expansion phase of the study, only patients with measurable disease will be enrolled. No anti-cancer therapies (inclusive of investigational therapies) are allowed 5 half-lives/4 weeks (whichever is longer) prior to study drug administration (6 weeks for nitrosoureas or mitomycin C).

ABI-011 will be administered via IV infusion for 30 minutes weekly on Days 1, 8, and 15 of a 28-Day cycle. The starting dose will be 2 mg/m2. Patients will be allowed to continue treatment until they experience progressive disease or unacceptable toxicity, withdraw consent, or their physician feels it is no longer in their best interest to continue on treatment.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following criteria to be enrolled in this study.

1. Patients ≥ 18 years of age (male and female).
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
3. Patients must be willing and able to sign an informed consent.
4. Cytologically or histologically confirmed solid tumor malignancy or lymphoma for which no curative standard approved therapy is available.
5. Patient agrees and is willing to provide 1 serial tumor biopsy (biopsies are mandatory), which would not put the patient or their treatment at significant risk.
6. During the dose-escalation phase, measurable or non-measurable disease as defined by RECIST criteria (Version 1.1); during the dose- expansion phase only; disease must be measurable by RECIST criteria (Version 1.1) (clinical or radiological).
7. Life expectancy of ≥ 12 weeks in the opinion of the investigator and medical monitor.
8. All adverse events (AEs) (except alopecia) of any prior chemotherapy, surgery, or radiotherapy must have resolved to Grade ≤ 1.
9. The following laboratory results must be present within the 14 days prior to the first administration of ABI-011:

   1. Hemoglobin ≥ 9 g/dL.
   2. Absolute neutrophil count (ANC) ≥1.5 x 109/L.
   3. Platelet count ≥ 100 x 109/L.
   4. Serum bilirubin ≤ 1.5 x upper limit of normal (ULN).
   5. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 ULN (except if liver metastases are present, then values must be ≤ 5 x ULN).
   6. Potassium, ionized calcium, and magnesium within normal limits (WNL).
   7. Creatine kinase WNL.
   8. Serum creatinine ≤ 1.5 x ULN.
   9. Activated partial thromboplastin time (aPTT) and prothrombin time (PT), or International Normal Ratio (INR) WNL.
   10. WNL levels of troponin I.
10. Women of child bearing potential and male patients who are not surgically sterile must be willing to practice contraceptive methods for the duration of the study and for 30-days following the last dose of study medication. Female patients must be postmenopausal (greater than 12 months from onset of menopause) or surgically sterile (have undergone bilateral oophorectomy or hysterectomy). Women of child bearing potential and women < 12 months since onset of menopause must agree to use an acceptable contraception method. If employing contraception, 2 of the following precautions must be used: vasectomy of partner, tubal ligation, vaginal diaphragm, intrauterine device, oral contraceptives (same oral contraceptive for a minimum of 3 months prior to screening), birth control injections, birth control implant, condom and spermicidal (gel/foam/cream/vaginal suppository). Male patients must be surgically sterile or agree to use a condom and acceptable contraception method with partner.
11. Women of childbearing potential and women < 12 months since onset of menopause must have a negative serum pregnancy test (ß-hCG) within 24 hours prior to the first administration of study drug

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study:

1. Inability to comply with study and follow-up procedures.
2. Women who are pregnant or breastfeeding (lactating).
3. Treatment with chemotherapy, hormonal therapy for cancer treatment (except leuprolide for prostate cancer), immunotherapy, biologic therapy, or radiation therapy as cancer therapy within 4 weeks or 5 half-lives, whichever is longer. Six weeks should have elapsed if prior chemotherapy treatment included nitrosoureas or mitomycin C.
4. Patients who have received antibody-based therapies within 28 days or 5 half-lives of the agent, whichever time period is longer.
5. Major surgery within 6 weeks before the first administration of study drug; needle aspirations, bone marrow biopsy and other similar procedures are allowable; minor surgery may be allowable following discussion and approval by Medical Monitor.
6. Prior treatment with tumor vascular disrupting agents (VDAs).
7. Any uncontrolled medical or psychiatric risk factors that would contraindicate the use or impair the ability of the patient to receive therapy per protocol or that may impose excessive risk to the patient.
8. Central nervous system (CNS) metastases. Patients who have a history of CNS metastases or who display signs or symptoms of CNS metastases should be imaged with magnetic resonance imaging (MRI) or computed tomography (CT) within 2 months of screening; if a patient has current symptoms, the MRI or CT should be performed at screening. Should active metastases be detected, these patients will not be enrolled. Patients with previously treated brain metastases will not be enrolled if taking steroids or anti-convulsants.
9. History of vascular neuropathy.
10. History of vasculitides (autoimmune or idiopathic).
11. History of retinopathy, including diabetic retinopathy. All patients must be evaluated by an ophthalmologist prior to study treatment.
12. Current use of medications that may cause corrected QT interval (QTc) prolongation. If the need to use these medications arises during the study, a discussion with and approval by the Medical Monitor is required.
13. History of allergy or hypersensitivity to any of the constituents of the ABI-011 formulation.
14. Active uncontrolled bacterial, viral, or fungal infection, requiring systemic therapy.
15. Known infection with human immunodeficiency virus (HIV) or known chronic active hepatitis B or hepatitis C virus (HBV/HCV) infection, unless a co-morbidity in patients with hepatocellular carcinoma (HCC).
16. Inability to be venipunctured and/or tolerate venous access.
17. Concurrent active second malignancy for which the patient is receiving therapy, excluding non-melanomatous skin cancer or carcinoma in situ of the cervix.
18. Patients requiring therapeutic anticoagulation (e.g. warfarin, low-molecular weight heparin, or other anticoagulant) or with history of any bleeding diathesis. Aspirin or low-dose warfarin for catheter maintenance is allowed.
19. Centrally-located lung tumors originating in the lungs and situated in the carinal bifurcation, the lung hila, or the main bronchi.
20. Cardiovascular exclusion criteria:

    1. Left Ventricular Ejection Fraction (LVEF) < 50% as measured by echocardiography.
    2. History (within prior 24 months) of either myocardial infarction or unstable or poorly controlled angina.
    3. Electrocardiogram findings suggestive of significant current or previous ischemic heart disease, or left bundle branch block.
    4. A cumulative doxorubicin dose of 550 mg/m2 or more; if patient has had radiation to the chest and the heart was in the radiation field the maximum cumulative doxorubicin dose is 300 mg/m².
    5. Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification.
    6. Congenital or acquired long QT syndrome.
    7. Uncontrolled hypertension: Blood pressure (BP) which when assessed on two different occasions (e.g. screening and baseline) is greater than 150 millimeters of mercury (mmHg) systolic and 90 mmHg diastolic despite receipt of antihypertensive medication.
    8. Any current or past history of clinically significant arrhythmias, including treatment with anti-arrhythmics.
    9. QTc prolongation defined as a QTc interval according to Bazett's formula of ≥ 450 msec for male patients or ≥470 msec for female patients at Baseline. Interval determination will be based on a mean value obtained from 3 sequential baseline electrocardiographs (ECGs) obtained at least 5 minutes apart.
    10. History of symptomatic peripheral vascular disease (venous or arterial) requiring surgical intervention or chronic therapy (other than aspirin).
21. Seizure disease requiring current anticonvulsant treatment.
22. History of previous head trauma, cerebrovascular accident or transient ischemic attack within 24 months of enrollment.
23. History of inflammatory bowel disease (active or past), or active peptic ulcer disease (prophylaxis with H2 blockers and proton pump inhibitors is acceptable).
24. History of previous, whole abdomen radiation therapy or Grade ≥ 1 residual toxicity from previous radiation therapy.
25. Administration of palliative radiotherapy for pain control within 7-days of planned administration of ABI-011.
26. Transfusion of blood products [red blood cells (RBC), white blood cells (WBC) or whole blood] or Hematopoietic growth factors or other hematologic support, such as erythropoiesis-stimulating agents, granulocyte-colony stimulating factor (G-CSF), or platelet transfusion(s) within 14 days of screening.
27. Participation in an investigational drug or device study within 30 days of screening for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-08-23 (Actual)

PRIMARY OUTCOMES:
Determine maximum tolerated dose (MTD) of ABI-011 | During Cycle 1 and each 28-Day treatment cycle, End of Study, Follow-up, approximately up to 1 year
  Determine the maximum tolerated dose (MTD) for repeated dosing of ABI-011

SECONDARY OUTCOMES:
Evaluate safety and toxicity profile of ABI-011 | During Cycle 1 and each 28-Day treatment cycle, End of Study, Follow-up, approximately up to 2 years total
  Evaluate safety and toxicity profile for repeated dosing of ABI-011. Number of subjects with adverse events (AEs), laboratory, electrocardiogram (ECG), echocardiogram, and ophthalmologic assessments, tumor pain and vital signs.
Evaluate pharmacokinetics (PK) analysis; elimination rate constant | Cycle 1 (Days 1,2,3); Cycle 2 (Days 1, 2, 3); Cycle 3 (Days 1, 2, 3)
  Evaluate drug concentration time data by individual subject for repeated dosing of ABI-011.
Evaluate pharmacokinetics (PK) analysis; elimination half-life | Cycle 1 (Days 1,2,3); Cycle 2 (Days 1, 2, 3); Cycle 3 (Days 1, 2, 3)
  Evaluate drug concentration time data by individual subject for repeated dosing of ABI-011.
Evaluate pharmacokinetics (PK) analysis; volume of distribution | Cycle 1 (Days 1,2,3); Cycle 2 (Days 1, 2, 3); Cycle 3 (Days 1, 2, 3)
  Evaluate drug concentration time data by individual subject for repeated dosing of ABI-011.
Evaluate pharmacokinetics (PK) analysis; maximum plasma drug concentration (Cmax) | Cycle 1 (Days 1,2,3); Cycle 2 (Days 1, 2, 3); Cycle 3 (Days 1, 2, 3)
  Evaluate drug concentration time data by individual subject for repeated dosing of ABI-011.
Evaluate pharmacokinetics (PK) analysis; time to maximum concentration (tmax) | Cycle 1 (Days 1,2,3); Cycle 2 (Days 1, 2, 3); Cycle 3 (Days 1, 2, 3)
  Evaluate drug concentration time data by individual subject for repeated dosing of ABI-011.
Evaluate pharmacokinetics (PK) analysis; area under the time-concentration curve (AUC) | Cycle 1 (Days 1,2,3); Cycle 2 (Days 1, 2, 3); Cycle 3 (Days 1, 2, 3)
  Evaluate drug concentration time data by individual subject for repeated dosing of ABI-011.
Tumor response | Baseline and Every 8 weeks through Cycle 6, then every 12 weeks, approximately up to 2 years total
  Tumor response based on assessment of target and non-target lesions according to response evaluation criteria in solid tumors (RECIST) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Mira Kistler, MD, Principal Investigator — Chan Soon-Shiong Institutes for Medicine
Locations (1):
- Chan Soon-Shiong Institute for Medicine, El Segundo, California, United States

IPD SHARING:
Plan to Share IPD: No